CLINICAL TRIAL: NCT04357210
Title: Uni-center, Retrospective Observational Study to Compare Outcomes of Fistulectomy With Primary Sphincteroplasty, Advancement Flap and Full-thickness Low Rectum Posterior Mobilization After Excision of a High Recurrent Anorectal Fistula
Brief Title: Anal Sphincter Reconstruction After High Recurrent Anorectal Fistula Excision
Status: Completed | Type: Observational
Sponsor: Russian Society of Colorectal Surgeons (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 76523
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Anorectal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- primary sphincteroplasty: end-to-end primary sphincteroplasty with interrupted sutures
  Interventions: Procedure: fistula tract excision and anal sphincter reconstruction
- muco-muscular advancement flap: A U-shaped muco-muscular flap was mobilized and fixed to the anoderm with one-row interrupted absorbable sutures
  Interventions: Procedure: fistula tract excision and anal sphincter reconstruction
- full-thickness low rectum posterior semicircular mobilization: Proximal parts of the internal sphincter and the longitudinal muscle were carefully separated from the underlying external sphincter and puborectalis muscle, moving further in the cranial direction, the Waldeyer's fascia was exposed and incised. Full-thickness posterior semicircular flap was fixed to anoderm
  Interventions: Procedure: fistula tract excision and anal sphincter reconstruction

INTERVENTIONS:
Procedure: fistula tract excision and anal sphincter reconstruction — The primary fistulous tract was excised together with any secondary tracts or residual cavities. Then on of the reconstructive steps was performed

SUMMARY:
A retrospective analysis of patients treated for recurrent posterior anorectal fistula, who previously had undergone radical excision of fistula-in-ano, was performed. Three types of surgical reconstruction were compared: fistulectomy with primary sphincteroplasty, muco-muscular advancement flap and full-thickness low rectum posterior semicircular mobilization.

DETAILED DESCRIPTION:
Radical surgical treatment of anorectal fistulas implies removal of the tract, which ideally should be followed by complete wound healing and good anal sphincter function. A big variety of techniques to restore the anal canal after fistula excision have been developed, however, none of them demonstrates excellent results in difficult clinical situations. Treatment of high anorectal fistulas, as well as recurrent fistulas, has always been the most challenging task even for expert colorectal surgeons, considering the need to safely restore the anal sphincters after surgical trauma in the presence of severe postoperative fibrosis and inflammatory changes.

In high recurrent anorectal fistulas, fistulotomy isn't a method of choice as division of a big portion of anal sphincter muscles leads to postoperative incontinence. Muco-muscular advancement flap is an accepted technique for the treatment of high transsphincteric fistulas, showing the best efficacy in unchanged anal canal. Whereas in recurrent disease, due to severe fibrotic deformation of the anal canal, creating an advancement flap can be technically difficult and lead to a complication high rate and postoperative incontinence.

Creation and safe fixation of an endorectal advancement flap (ERAF) in the setting of postoperative fibrosis and perifistular inflammation can be technically difficult. Thus, mobilizing a full-thickness flap is preferred.

After coring out a high transsphincteric or suprasphincteric fistula, the wound from the inside of the anal canal is located close to the anorectal junction, where internal and external anal sphincter fuse with the levator ani muscles. When a full-thickness ERAF is created in this situation, first the surgeon enters the intersphincteric plane, and upward dissection brings him straight to the supralevator space.

This maneuver has much in common with mobilising the distal part of rectum as a part of intersphincteric resections or transanal mesorectal excision for rectal cancer [35] , [36] . After the upper part of the rectum has been mobilized, a surgeon from the perineal team makes a circular incision of the anal canal above the dentate line, enters the intersphincteric space and continues dissection in cranial direction following the surface of the mesorectal fascia, thus separating the lower part of mesorectum from the levator ani muscles.

Being an expert in intersphincteric resections, the leading surgeon utilized this approach in three patients after excision of a high recurrent anal fistula. Sphincteroplasty and standard ERAF creation were not possible due to severe fibrosis, so mobilizing the posterior semicircle of the rectum the same way as in intersphincteric rectal resection was deemed to be the last resort in order to close the wound. In fact, a wide well-vascularized posterior ERAF was created. The upward dissection was continued until the Waldeyer's septum was reached and divided to ensure tension-free fixation of the flap in the anal canal.

ELIGIBILITY:
Inclusion Criteria:

* recurrent posterior anorectal fistula
* previously had undergone radical excision
* contrast-enhanced MRI performed preoperatively
* colonoscopy preoperatively

Exclusion Criteria:

* Crohn's disease
* superficial fistulas
* low intersphincteric fistulas
* infections (anorectal sepsis, tuberculosis, HIV)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with high recurrent posteriorly located anorectal fistulas
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 12 months
  The rate of any symptoms or clinical signs related to recurrence of anorectal fistula: persistent non-healing wound, discharge through the postoperative scar after complete wound healing or an abscess in operation area confirmed with ultrasound or MRI

SECONDARY OUTCOMES:
Operative time | Day 0
  Duration of the operation in minutes
Intraoperative blood loss | Day 0
  The volume of blood lost in the course of the procedure
Pain intensity | postoperative days 1, 3, 7, 14, 28
  The intensity of pain as measured with Visual Analogue Scale (VAS) having 10 grades, with 0 representing no pain and 10 representing the most intensive pain that a person can tolerate.
Anal incontinence score | postoperative days 1, 3, 7, 14, 28
  Evaluated with Cleveland Clinic Florida Fecal Incontinence (CCFFI) score that has 5 questions with 0 to 4 scores assigned to each of them. The total score is calculated, and 0 is referred as no incontinence and 20 - complete incontinence.
Complete wound healing time | 1 year
  The time period between the procedure and the date when complete wound healing was confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Study Director — Director

IPD SHARING:
Plan to Share IPD: Undecided
fistula tract location, wound size, depth, the presence of exudate, complete/incomplete healing, presence of anal incontinence, fistula recurrence, any complications.